CLINICAL TRIAL: NCT07130344
Title: PERCIST Evaluation of Trastuzumab Deruxtecan in the Treatment of HER2 Low Breast Cancer
Acronym: PERPETUAL
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Paul Strauss (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2024-008
Record Dates: First submitted 2025-08-12; First posted 2025-08-19 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Metastatic Breast Cancer; HER 2 Low-expressing Breast Cancer
Keywords: Breast Cancer; 18F-FDG PET-CT; T-DXd
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SOC arm (Active Comparator): Patient will be followed by TAP CT-scan and bone scintigraphy every 3 months, until progression or new treatment initiation or until 2 years whichever occurs first.
  Interventions: Procedure: TAP CT-scan; Procedure: Bone scintigraphy
- Experimental arm (Experimental): Patient will be followed by 18F-FDG PET-CT every 3 months, until progression or new treatment initiation or until 2 years whichever occurs first.
  Interventions: Procedure: 18F-FDG PET-CT

INTERVENTIONS:
Procedure: TAP CT-scan — Patient in the SOC arm will be followed by TAP CT-scan every 3 months, until progression or new treatment initiation or until 2 years whichever occurs first.
  Arms: SOC arm
Procedure: Bone scintigraphy — Patient in the SOC arm will be followed by bone scintigraphy every 3 months, until progression or new treatment initiation or until 2 years whichever occurs first.
  Arms: SOC arm
Procedure: 18F-FDG PET-CT — Patient in the experimental arm will be followed by 18F-FDG PET-CT every 3 months, until progression or new treatment initiation or until 2 years whichever occurs first.
  Arms: Experimental arm

SUMMARY:
The development of trastuzumab deruxtecan (T-DXd), an anti-HER2 conjugated antibody, has changed the therapeutic landscape of breast cancer. Anti-HER2 molecules were previously used exclusively in cases of HER2-positive breast cancer (IHC HER2 3+ or HER2 2+ with amplified FISH/SISH).

Since a couple of years, T-DXd is becoming a reference treatment in patients with low HER2 breast cancer (IHC 1+ or 2+ with non-amplified FISH/SISH) after hormone therapy and at least one line of chemotherapy. The results of the DB04 trial revealed that T-DXd increased progression-free survival and overall survival compared to investigator's choice chemotherapy, in HER2 low breast cancers patients after one or two previous lines of chemotherapy (Modi, S. et al., 2022).

In several trials, T-DXd validation was done thanks to radiological evaluation based on conventional imaging, computed tomography scan (CT-scan) with or without contrast dye injection and bone scintigraphy.

18F-Fluorodeoxyglucose positron emission tomography coupled with computed tomography (18F-FDG PET-CT) represents a major tool for diagnosis, staging, and therapeutic follow-up in oncology.

It was demonstrated that 18F-FDG PET-CT is more sensitive in detecting metastatic disease progression in HER2-positive breast cancer patients treated with trastuzumab and pertuzumab or trastuzumab and lapatinib (Ma, G. et al., 2023 et Lin, N. U. et al., 2015). Moreover, a prospective study investigated the correlation between the response rate defined by 18F-FDG PET-CT and thoraco-abdomino-pelvic CT-scan (TAP CT-scan) and the progression-free survival of patients with breast cancer. PET evaluation allowed better identification of responders versus non-responders, with a significant correlation with progression-free survival (Vogsen, M. et al., 2023).

With this study, the investigators aim to determine the role of 18F-FDG PET-CT in evaluating T-DXd treatment in patients with metastatic low HER2 breast cancer. 18F-FDG PET-CT could be an earlier evaluation tool than CT-scan in identifying non-responsive patients; and thus, avoid continuing an expensive treatment with an unfavorable toxicity profile, which could worsen both patient prognosis and quality of life.

DETAILED DESCRIPTION:
Screening period will last 28 days. Each participant will have baseline evaluation by TAP CT-scan, bone scintigraphy and 18F-FDG PET-CT.

After randomization, patient will start T-DXd treatment according to SOC until progression or toxicity. Patient will be followed by TAP CT-scan and bone scintigraphy (SOC arm) or 18F-FDG PET-CT (experimental arm) every 3 months, until progression or new treatment initiation or death or until 2 years whichever occurs first.

ELIGIBILITY:
Inclusion Criteria:

1. Age greater than or equal to 18 years at inclusion
2. Cytological or histological confirmation of the diagnosis of low HER2 breast cancer (IHC 1+ or 2+ with non-amplified FISH/SIS)
3. Metastatic disease according to RECIST 1.1
4. Indication of T-DXd treatment
5. Patient (male or female of childbearing potential) using a highly effective contraceptive method
6. Women of childbearing potential must have a negative pregnancy test within 72 hours before starting treatment
7. Willingness and ability to comply with the visit schedule, treatment regimens, examinations and other procedures planned in the study
8. Patient enrolled in a health insurance plan or beneficiary of such a plan
9. Signed informed consent obtained before inclusion (after giving clear, fair and appropriate information)

Exclusion Criteria:

1. Allergy to contrast dye
2. Contra-indication to PET-CT
3. Any active infection or uncontrolled intercurrent pathology
4. Patient with a life expectancy lower than 3 months
5. Ongoing participation in another clinical trial with an investigational treatment
6. Pregnant or breastfeeding women
7. Persons deprived of their freedom or under guardianship or incapable of giving consent
8. Any psychiatric illness/social situation that may limit compliance with study procedures or prevent the patient from giving written informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 262 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2028-12 (Estimated); Study Completion 2030-09 (Estimated)

PRIMARY OUTCOMES:
Objective response rate | at 3 months
  Radiological response according to PERCIST 1.0 criteria in experimental arm and RECIST 1.1 criteria in SOC arm. Number of patients who had an objective response at 3 months in both arms. The evaluation is carried out by the investigator.

SECONDARY OUTCOMES:
Progression-free survival | Every 3 months until the date of first documented progression or new therapy initiation or date of death or until 2 years, whichever occurs first.
  Progression events will be collected (progression according to PERCIST 1.0 criteria in experimental arm and RECIST 1.1 criteria in SOC arm or death whatever the cause).
Time until new therapy initiation | Until initiation of a new therapy or until 2 years, whichever occurs first.
  Time from inclusion to initiation of new therapy.
Overall survival | From date of inclusion until the date of death or lost to follow-up or until 2 years, whichever occurs first.
  The patient's condition (alive, deceased from whatever cause or lost to follow-up) will be collected. Patients alive at the time of analysis will be censored on the date of last contact.
Response duration | Every 3 months until the date of first documented progression or new therapy initiation or date of death or until 2 years, whichever occurs first.
  Time from date of first documented response (complete or partial response) to date of first subsequent progression or death from any cause.
Patient Quality of life | Every 3 months until the date of first documented progression or new therapy initiation or date of death or until 2 years, whichever occurs first.
  Assessment of all dimensions of the European Organization for Research and Treatment of Cancer (EORTC) QLG Core Questionnaire (EORTC QLQ-C30). Difference on specific symptom scales (from 1 = " not at all " to 4 = " very much ", or from 1 = " really bad " to 7 = " excellent ").

CONTACTS AND LOCATIONS:
Overall Officials: François SOMME, Principal Investigator — Institut de cancérologie Strasbourg Europe
Locations (1):
- ICANS, Strasbourg, France